CLINICAL TRIAL: NCT00949897
Title: A Randomized, Prospective, Controlled Trial for Lateral Column Lengthening in Adult Acquired Flatfoot Using Biofoam Porous Metal Compared With Allograft
Brief Title: Comparison Study of Biofoam Porous Metal Versus Allograft to Treat Adult Acquired Flatfoot
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding terminated
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Collaborators: Stryker Trauma and Extremities (Industry)
Responsible Party: Anne J. Schwoebel, Executive Director, OrthoCarolina Research Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120813B
Record Dates: First submitted 2009-07-29; First posted 2009-07-31 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Adult Acquired Flatfoot
Keywords: Adult Acquired Flatfoot; Biofoam Porous Metal Implant; Allograft Bone Wedge

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biofoam (Active Comparator)
  Interventions: Device: Biofoam
- Iliac Crest Allograft with locked plate (Active Comparator)
  Interventions: Other: Iliac Crest Allograft with locked plate

INTERVENTIONS:
Device: Biofoam — Device
  Other Names: 510(k) Number: K073535
  Arms: Biofoam
Other: Iliac Crest Allograft with locked plate
  Other Names: Iliac Crest Allograft
  Arms: Iliac Crest Allograft with locked plate

SUMMARY:
The purpose of this study is to compare the clinical and radiographic outcomes of a randomized, consecutive series of adult patients, with an acquired flatfoot, treated with a lateral column lengthening using an allograft bone wedge versus a titanium porous metal implant (Biofoam, Wright Medical).

Null hypothesis: At six months postoperatively, there is no difference in the degree of correction as measured by the talonavicular coverage angle between patients randomized to allograft and Biofoam.

Alternative hypothesis: At six months postoperatively, the degree of correction as measured by the talonavicular coverage angle will be less in patients randomized to allograft than the degree of correction in patients randomized to Biofoam.

ELIGIBILITY:
Inclusion Criteria:

* Ages 25-75
* Unresponsive to conservative treatment
* Patient with acquired flatfoot deformity, who is a candidate for lateral column lengthening (Stage IIB) = (greater than > 40% uncoverage of talar head by navicular on standing AP radiograph)

Exclusion Criteria:

* Less than 25 years of age and greater than 75 years
* Pre-existing infection
* Peripheral neuropathy
* Charcot arthropathy
* Peripheral vascular disease
* Rhematoid Arthritis (RA) or inflammatory arthropathy
* Metal allergy or sensitivity to metal

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The degree of correction as measured by talonavicular coverage angle, which is used to quantify the degree of deformity. Degree of correction is defined as the difference between the preoperative and postoperative talonavicular coverage angle. | 2 weeks, 6 weeks, 12 weeks, and 6 months

SECONDARY OUTCOMES:
American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Score | 2 weeks, 6 weeks, 3 months, and 6 months
Foot Function Index (FFI) Score | 2 weeks, 6 weeks, 3 months, and 6 months
Pain Visual Analog Scale (VAS) | 2 weeks, 6 weeks, 3 months, and 6 months
Implant failure | 2 weeks, 6 weeks, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Anderson, MD, Principal Investigator — OrthoCarolina, P.A.
Locations (1):
- OrthoCarolina, P.A., Charlotte, North Carolina, United States